CLINICAL TRIAL: NCT04549766
Title: The Predictive Value of PRECISE DAPT Score in Patients With ST Segment Elevation Myocardial Infarction (STEMI) After Primary Percutaneous Coronary Intervention (PPCI)
Brief Title: Predictive Value of PRECISE DAPT Score in STEMI Patients After Primary PCI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Madona Atef, Doctor, Assiut University
Other Study IDs: PRECISE DAPT score
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI)
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: calculate PRECISE DAPT score using clinical data — calculate PRECISE DAPT score using clinical data in STEMI patients after PPCI

SUMMARY:
To investigate the predictive value of PRECISE DAPT score in relation to coronary slow flow & other short term major adverse cardiovascular events (MACE) post PPCI .

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the leading cause of death around the world and more than 4 million people die every year due to CAD in Europe.[1] The incidence of ST elevation myocardial infarction (STEMI) appears to be declining; however, it is still an important issue in cardiovascular medicine.[2] Initial risk assessment is important for STEMI to estimate adverse cardiovascular outcomes. Previous studies demonstrated that increased age, advanced Killip class, heart rate, arterial hypotension, increased serum creatinine, white blood cell counts, and hemoglobin levels were predictors of in-hospital and early mortality in patients with STEMI treated with primary percutaneous coronary intervention (PPCI).[3,4 ]Therefore, risk scores including the aforementioned parameters were developed to estimate mortality in patients with STEMI.

No-reflow is still a challenging major issue in the management of the patients with STEMI undergoing primary PCI. It is defined as inadequate myocardial perfusionthrough a given segment of the coronary circulation without angiographic evidence of mechanical vessel obstructionas [5] Angiographic no-reflow defined as less than Thrombolysis In Myocardial Infarction (TIMI) 3 flow [6] and angiographic success was defined as TIMI Grade 3 Flow .

PRECISE-DAPT score includes age, creatinine clearance, white blood cell counts, hemoglobin levels, and prior spontaneous bleeding [7]. All these factors have a close relationship with coronary artery disease (CAD) and complications [8-10]. Therefore, in this study, we aimed to evaluate the association of admission PRECISE-DAPT score with the development of slow flow & bleeding & othershort term cardiovascular complications that develop in patients with STEMI treated with primary PCI.

ELIGIBILITY:
Inclusion Criteria:1.Subjects diagnosed as STEMI accordind to fourth universal definition with age range from 18 to 75 years underwent PPCI at cardiology hospital assiut university hospital.[11].

2..Patients elegable for PPCI with STEMI within 12 h of symptom onset, provided it can be performed expeditiously (i.e. 120 min from STEMI diagnosis)[12]

-

Exclusion Criteria:1-late presentation with STEMI more than 12 hr & door to ballon more than 120 min including rescue PCI .

2- cardiogenic shock 3-Patients known to have autoimmune disease (e.g vasculitis ) 4- platelate count less than 100000 IU . 5- prothrombin concentration less than 60% 6- Patients taking triple anti thrombotics .

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed as STEMI accordind to fourth universal definition with age range from 18 to 75 years underwent PPCI at cardiology hospital assiut university hospital eligible for PPCI with STEMI within 12 h of symptom onset, provided it can be performed expeditiously (i.e. 120 min from STEMI diagnosis)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Follow up complications after PPCI | 3 months
  calculating PRECISE DAPT score and follow up patients for three months whether these complications as coronary slow flow &primary MACE &secondary MACE &bleeding

SECONDARY OUTCOMES:
Predictive value of PRECISE DAPT score | 3 months
  Whether there is relation between PRECISE DAPT score &post PPCI short term complications or not

CONTACTS AND LOCATIONS:
Overall Officials: Aly Mohamed, Lecturer, Principal Investigator — Assiut University

REFERENCES:
- [Background] Townsend N, Wilson L, Bhatnagar P, Wickramasinghe K, Rayner M, Nichols M. Cardiovascular disease in Europe: epidemiological update 2016. Eur Heart J. 2016 Nov 7;37(42):3232-3245. doi: 10.1093/eurheartj/ehw334. Epub 2016 Aug 14. No abstract available. PMID 27523477
- [Background] Widimsky P, Wijns W, Fajadet J, de Belder M, Knot J, Aaberge L, Andrikopoulos G, Baz JA, Betriu A, Claeys M, Danchin N, Djambazov S, Erne P, Hartikainen J, Huber K, Kala P, Klinceva M, Kristensen SD, Ludman P, Ferre JM, Merkely B, Milicic D, Morais J, Noc M, Opolski G, Ostojic M, Radovanovic D, De Servi S, Stenestrand U, Studencan M, Tubaro M, Vasiljevic Z, Weidinger F, Witkowski A, Zeymer U; European Association for Percutaneous Cardiovascular Interventions. Reperfusion therapy for ST elevation acute myocardial infarction in Europe: description of the current situation in 30 countries. Eur Heart J. 2010 Apr;31(8):943-57. doi: 10.1093/eurheartj/ehp492. Epub 2009 Nov 19. PMID 19933242
- [Background] Yusufali A, Zubaid M, Al-Zakwani I, Alsheikh-Ali AA, Al-Mallah MH, Al Suwaidi J, AlMahmeed W, Rashed W, Sulaiman K, Amin H. Validation of the GRACE Risk score for hospital mortality in patients with acute coronary syndrome in the Arab Middle East. Angiology. 2011 Jul;62(5):390-6. doi: 10.1177/0003319710387921. Epub 2011 Feb 8. PMID 21307002
- [Background] Puymirat E, Simon T, Steg PG, Schiele F, Gueret P, Blanchard D, Khalife K, Goldstein P, Cattan S, Vaur L, Cambou JP, Ferrieres J, Danchin N; USIK USIC 2000 Investigators; FAST MI Investigators. Association of changes in clinical characteristics and management with improvement in survival among patients with ST-elevation myocardial infarction. JAMA. 2012 Sep 12;308(10):998-1006. doi: 10.1001/2012.jama.11348. PMID 22928184
- [Background] Kloner RA, Ganote CE, Jennings RB. The "no-reflow" phenomenon after temporary coronary occlusion in the dog. J Clin Invest. 1974 Dec;54(6):1496-508. doi: 10.1172/JCI107898. PMID 4140198
- [Background] Abbo KM, Dooris M, Glazier S, O'Neill WW, Byrd D, Grines CL, Safian RD. Features and outcome of no-reflow after percutaneous coronary intervention. Am J Cardiol. 1995 Apr 15;75(12):778-82. doi: 10.1016/s0002-9149(99)80410-x. PMID 7717278
- [Background] Costa F, van Klaveren D, James S, Heg D, Raber L, Feres F, Pilgrim T, Hong MK, Kim HS, Colombo A, Steg PG, Zanchin T, Palmerini T, Wallentin L, Bhatt DL, Stone GW, Windecker S, Steyerberg EW, Valgimigli M; PRECISE-DAPT Study Investigators. Derivation and validation of the predicting bleeding complications in patients undergoing stent implantation and subsequent dual antiplatelet therapy (PRECISE-DAPT) score: a pooled analysis of individual-patient datasets from clinical trials. Lancet. 2017 Mar 11;389(10073):1025-1034. doi: 10.1016/S0140-6736(17)30397-5. PMID 28290994
- [Background] Zeidman A, Fradin Z, Blecher A, Oster HS, Avrahami Y, Mittelman M. Anemia as a risk factor for ischemic heart disease. Isr Med Assoc J. 2004 Jan;6(1):16-8. PMID 14740503
- [Background] Mehta RH, Starr AZ, Lopes RD, Hochman JS, Widimsky P, Pieper KS, Armstrong PW, Granger CB; APEX AMI Investigators. Incidence of and outcomes associated with ventricular tachycardia or fibrillation in patients undergoing primary percutaneous coronary intervention. JAMA. 2009 May 6;301(17):1779-89. doi: 10.1001/jama.2009.600. PMID 19417195
- [Background] Chatterjee S, Chandra P, Guha G, Kalra V, Chakraborty A, Frankel R, Shani J. Pre-procedural Elevated White Blood Cell Count and Neutrophil-Lymphocyte (N/L) Ratio are Predictors of Ventricular Arrhythmias During Percutaneous Coronary Intervention. Cardiovasc Hematol Disord Drug Targets. 2011;11(2):58-60. doi: 10.2174/187152911798346981. PMID 22044033
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Thiemann DR, Coresh J, Oetgen WJ, Powe NR. The association between hospital volume and survival after acute myocardial infarction in elderly patients. N Engl J Med. 1999 May 27;340(21):1640-8. doi: 10.1056/NEJM199905273402106. PMID 10341277
- [Background] Valgimigli M, Bueno H, Byrne RA, Collet JP, Costa F, Jeppsson A, Juni P, Kastrati A, Kolh P, Mauri L, Montalescot G, Neumann FJ, Petricevic M, Roffi M, Steg PG, Windecker S, Zamorano JL, Levine GN; ESC Scientific Document Group; ESC Committee for Practice Guidelines (CPG); ESC National Cardiac Societies. 2017 ESC focused update on dual antiplatelet therapy in coronary artery disease developed in collaboration with EACTS: The Task Force for dual antiplatelet therapy in coronary artery disease of the European Society of Cardiology (ESC) and of the European Association for Cardio-Thoracic Surgery (EACTS). Eur Heart J. 2018 Jan 14;39(3):213-260. doi: 10.1093/eurheartj/ehx419. No abstract available. PMID 28886622
- [Background] 14-TIMI Flow Grade is scored from 0 to 3. It is a powerful predictor of outcome. Here shown are the findings from the TIMI 1 trial. TIMI, Thrombolysis in Myocardial Infarction. [Data from Flyngenring BP, Sheehan FH, Kennedy JW, Dodge HT, Braunwald E. Does arterial patency 90 minutes following thrombolytic therapy predict 42 day survival? J Am Coll Cardiol. 1991;17(Suppl A):275A.]
- [Background] 15- Gibson CM, Cannon CP, Daley WL; et al. (1996).
- [Background] 16 Gibson CM, Murphy SA, Rizzo MJ; et al. (1999).
- [Background] 17 - Gibson CM, Cannon CP, Murphy SA, Marble SJ, Barron HV, Braunwald E (2002).
- [Background] 18- January 2012Cardiology International 13(3):98-101
- [Background] 19-de Jong M, van der Worp HB, van der Graaf Y, Visseren FL, Westerink J (2017).
- [Background] Arnott C, Li Q, Kang A, Neuen BL, Bompoint S, Lam CSP, Rodgers A, Mahaffey KW, Cannon CP, Perkovic V, Jardine MJ, Neal B. Sodium-Glucose Cotransporter 2 Inhibition for the Prevention of Cardiovascular Events in Patients With Type 2 Diabetes Mellitus: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2020 Feb 4;9(3):e014908. doi: 10.1161/JAHA.119.014908. Epub 2020 Jan 29. PMID 31992158
- [Background] Ndrepepa G, Schuster T, Hadamitzky M, Byrne RA, Mehilli J, Neumann FJ, Richardt G, Schulz S, Laugwitz KL, Massberg S, Schomig A, Kastrati A. Validation of the Bleeding Academic Research Consortium definition of bleeding in patients with coronary artery disease undergoing percutaneous coronary intervention. Circulation. 2012 Mar 20;125(11):1424-31. doi: 10.1161/CIRCULATIONAHA.111.060871. Epub 2012 Feb 17. PMID 22344040